CLINICAL TRIAL: NCT03498170
Title: An Open-label, 2-period, Single-sequence, Crossover Study to Evaluate the Effect of Multiple Oral Dosing of Itraconazole on BCT197 Systemic Exposure in Healthy Male Participants
Brief Title: The Effect of Itraconazole on BCT197 Exposure in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mereo BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MBCT103
Record Dates: First submitted 2018-04-06; First posted 2018-04-13 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-04

CONDITIONS: Interaction
Keywords: Healthy Male Volunteers
MeSH Terms: interventions — acumapimod; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Period 1 and Period 2 (Other): Period 1 - BCT197 14mg on Day 1
  Period 2 - itraconazole 200mg on Day 1 to 14 and BCT197 14mg on Day 7
  Interventions: Drug: BCT197; Drug: Itraconazole 200 mg

INTERVENTIONS:
Drug: BCT197 — Single dose of BCT197
  Other Names: Acumapimod
Drug: Itraconazole 200 mg — Single dose of itraconazole
  Other Names: Sporanox

SUMMARY:
An Open-label, 2-period, Single-sequence, Crossover Study to Evaluate the Effect of Multiple Oral Dosing of Itraconazole on BCT197 Systemic Exposure in Healthy Male Participants.

DETAILED DESCRIPTION:
This will be an open label study conducted in healthy male participants at a single centre. Each participant will participate in a screening visit and 2 study periods. At the first study period, all participants will receive a single dose of BCT197 and at study period 2, all participants will receive 14 daily doses of itraconazole and a single dose of BCT197.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male participants.
* Non-smokers (including e-cigarettes).
* Body mass index (BMI) ≥ 18 and ≤ 30 kg/m2.
* Willing to use highly effective barrier contraception methods.
* Male participants must not donate sperm during the study.

Exclusion Criteria:

* Any participants with pre-existing active skin disease.
* Laboratory values at screening which are deemed to be clinically significant.
* Participants with abnormal liver function tests.
* 12 Lead ECG with QTcF >450 msec.
* Allergy to any of BCT197 excipients.
* Known hypersensitivity or intolerance to itraconazole.
* Taking medications known to cause QTc prolongation.
* Positive for human immunodeficiency virus (HIV), hepatitis B or hepatitis C.
* Any clinically significant illness within 30 days prior to study drug administration.
* Participants who, in the opinion of the Investigator, are unsuitable for participation in the study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2018-05-09 (Actual)

PRIMARY OUTCOMES:
Maximum Measurable Plasma Concentration (Cmax) BCT197 in the presence and absence of itraconazole. | Pre-dose to Day 15
  Period 1: Pre-dose and 1, 2, 4, 6, 12, 24, 36, 48, 72, 96, 144 and 168 hours post BCT197 dose on Day 1.
  Period 2: Pre-dose and 1, 2, 4, 6, 12, 24, 36, 48, 72, 96, 144, 168 and 192 hours post BCT197 dose on Day 7.
Area under the plasma concentration-time curve (AUC) BCT197 in the presence and absence of itraconazole. | Pre-dose to Day 15
  Period 1: Pre-dose and 1, 2, 4, 6, 12, 24, 36, 48, 72, 96, 144 and 168 hours post BCT197 dose on Day 1.
  Period 2: Pre-dose and 1, 2, 4, 6, 12, 24, 36, 48, 72, 96, 144, 168 and 192 hours post BCT197 dose on Day 7.

SECONDARY OUTCOMES:
The number of adverse events during administration of BCT197 alone and in the presence of itraconazole. | Day 1 to Day 21

OTHER OUTCOMES:
Corrected QT interval of the electrocardiogram (QTc). | Pre-dose to Day 15
  Period 1: Pre-dose, 2, 4, 6, 8, 24 and 168 hours post BCT197 dose on Day 1. Period 2: Pre-dose, 2, 4, 6, 8, 24, 168 and 192 hours post BCT197 dose on Day 7.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Parkin, PhD FRCP, Study Director — Mereo BioPharma
Locations (1):
- inVentiv Health Clinical Research Services LLC, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No